CLINICAL TRIAL: NCT01898338
Title: Randomized Multicenter Study to Assess Efficacy of Daptomycin Plus Fosfomycin Versus Daptomycin Monotherapy for Treatment of Methicillin Resistant Staphylococcus Aureus Bacteremia in Hospitalized Patients
Brief Title: Efficacy of Daptomycin Plus Fosfomycin Versus Daptomycin for Treatment of MRSA Bacteremia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Miquel Pujol (Other)
Collaborators: Hospital Universitari de Bellvitge (Other)
Responsible Party: Sponsor-Investigator, Miquel Pujol, MD and PhD, Spanish Network for Research in Infectious Diseases
Organization: Spanish Network for Research in Infectious Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BACSARM; 2013-000586-37 (EudraCT Number)
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Staph Aureus Methicillin Resistant Bacteremia
Keywords: MRSA; bacteremia; therapy
MeSH Terms: conditions — Bacteremia | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fosfomycin and Daptomycin (Experimental): fosfomycin 2gr/6h + 10mg/kg/24h iv during 14 or 28 days
  Interventions: Drug: Fosfomycin 2gr/6h iv; Drug: Daptomycin 10mg/kg/24h iv
- Daptomycin (Active Comparator): daptomycin 10mg/kg/cada 24h iv during 14 or 28 days
  Interventions: Drug: Fosfomycin 2gr/6h iv

INTERVENTIONS:
Drug: Fosfomycin 2gr/6h iv
Drug: Daptomycin 10mg/kg/24h iv
  Arms: Fosfomycin and Daptomycin

SUMMARY:
To demonstrate that the combination of daptomycin and fosfomycin is superior to daptomycin alone in the treatment of methicillin resistant Staphylococcus aureus (MRSA) bacteremia.

DETAILED DESCRIPTION:
The mortality associated to MRSA bacteremia remains higher than 30% of episodes despite the availability of new antibiotics. Objective: To demonstrate that the combination of daptomycin and fosfomycin is superior to daptomycin alone in the treatment of methicillin resistant Staphylococcus aureus (MRSA) bacteremia. Design: Randomized, open-label and multicenter study. Intervention: Patients with MRSA bacteremia will be randomized (1:1) in Group 1: daptomycin 10mg/Kg/24h intravenous (iv) and Group 2: daptomycin 10 mg/kg/24 iv plus fosfomycin and 2g/6h iv. Duration of therapy will be 10-14 days for uncomplicated bacteremia and up to 42 days for complicated bacteremia. Follow up: There will be a clinical and microbiological evaluation at baseline, during treatment and at week 6 after the end of therapy (test of cure visit, TOC). Complicated bacteremia was considered if: a) persistence of a positive blood culture at 72-96 h from the start of antibiotic, b) evidence of spread of infection (metastatic infection) c) infection involving a non-removable device in less than 4 days. Sample size: Assuming 60% cure rate with daptomycin and a 20% difference in cure rates between both groups, we estimated that 103 patients will be needed for each group (α:0.05, ß: 0.2). Main endpoint: clinical and microbiological response at the TOC visit. Treatment success was defined as the resolution of clinical signs and symptoms and negative blood culture. Treatment failure was defined if any of the following situations: a) lack of clinical response at 72 h or more after initiation of the study therapy b) persistent bacteremia (positive blood culture on day 7 after randomization), c) withdrawal of treatment due to adverse effects or for any other reason based on clinical judgment. d) relapse of MRSA bacteremia before the TOC visit e) death for any reason before the TOC visit. Secondary endpoints: evaluation in both groups of clinical and microbiological response at end of therapy (EOT visit); mortality at EOT and TOC visit; persistent MRSA bacteremia; recurrence of MRSA bacteremia (positive blood culture when previous ones were negative); emergence of daptomycin or fosfomycin resistance and severe adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 1 positive blood culture to MRSA within 72h up to randomization
* Adult patients, equal or older than 18 years old
* Signed informed consent
* Mandatory use of contraception methods for fertile women during the study period and for 6 months after stopping antibiotic therapy

Exclusion Criteria:

* Polymicrobial bacteremia
* Pneumonia associated to the bacteremia
* Severe clinical status with expected survival of less than 24 hours
* Allergy to daptomycin or fosfomycin
* A positive pregnancy test at the time of inclusion
* Any clinical condition that requires additional antibiotic therapy with microbiological activity against MRSA
* Patient already included in another clinical trial
* Prior history of eosinophilic pneumonia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2013-12; Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Therapy response | at week 6 after end of therapy (an average of 8 to 12 weeks from the beginnig of therapy)
  Therapy response is considered if clinical and microbiological response is achieved at week 6 after end of therapy

SECONDARY OUTCOMES:
Mortality | participants will be followed an average of 8 to 12 weeks from the begining of therapy
Severe adverse effects | participants will be followed an average of 8 to 12 weeks from the begining of therapy
  whatever
Number of persistent bacteremia | participants will be followed an average of 8 to 12 weeks from the begining of therapy
  Defined as a positive blood culture on day 7 after starting the study therapy
Bacteremia recurrence | participants will be followed an average of 8 to 12 weeks from the begining of therapy
  Defined as a positive blood culture to MRSA when previous ones were negative
Therapy response at end of therapy (EOT visit) | at end of therapy
  Success is considered if clinical resolution and negative blood culture at end of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Pujol, MD, PhD, Study Director — (Infectious Diseases Service) Hospital Universitari de Bellvitge
Locations (18):
- Spain (18):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Universitari Mútua de Terrassa, Terrassa, Barcelona
  - Hospital de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital del Mar- Parc de Salut Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital General Gregorio Marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Asistencial Son Espases, Palma de Mallorca
  - Hospital Virgen Macarena, Seville
  - Hospital Universitari Joan XXIII, Tarragona

REFERENCES:
- [Background] Cosgrove SE, Sakoulas G, Perencevich EN, Schwaber MJ, Karchmer AW, Carmeli Y. Comparison of mortality associated with methicillin-resistant and methicillin-susceptible Staphylococcus aureus bacteremia: a meta-analysis. Clin Infect Dis. 2003 Jan 1;36(1):53-9. doi: 10.1086/345476. Epub 2002 Dec 13. PMID 12491202
- [Background] Chang FY, Peacock JE Jr, Musher DM, Triplett P, MacDonald BB, Mylotte JM, O'Donnell A, Wagener MM, Yu VL. Staphylococcus aureus bacteremia: recurrence and the impact of antibiotic treatment in a prospective multicenter study. Medicine (Baltimore). 2003 Sep;82(5):333-9. doi: 10.1097/01.md.0000091184.93122.09. PMID 14530782
- [Background] Fowler VG Jr, Boucher HW, Corey GR, Abrutyn E, Karchmer AW, Rupp ME, Levine DP, Chambers HF, Tally FP, Vigliani GA, Cabell CH, Link AS, DeMeyer I, Filler SG, Zervos M, Cook P, Parsonnet J, Bernstein JM, Price CS, Forrest GN, Fatkenheuer G, Gareca M, Rehm SJ, Brodt HR, Tice A, Cosgrove SE; S. aureus Endocarditis and Bacteremia Study Group. Daptomycin versus standard therapy for bacteremia and endocarditis caused by Staphylococcus aureus. N Engl J Med. 2006 Aug 17;355(7):653-65. doi: 10.1056/NEJMoa053783. PMID 16914701
- [Background] Rehm SJ, Boucher H, Levine D, Campion M, Eisenstein BI, Vigliani GA, Corey GR, Abrutyn E. Daptomycin versus vancomycin plus gentamicin for treatment of bacteraemia and endocarditis due to Staphylococcus aureus: subset analysis of patients infected with methicillin-resistant isolates. J Antimicrob Chemother. 2008 Dec;62(6):1413-21. doi: 10.1093/jac/dkn372. Epub 2008 Sep 8. PMID 18782781
- [Background] Gudiol F, Aguado JM, Pascual A, Pujol M, Almirante B, Miro JM, Cercenado E, Dominguez Mde L, Soriano A, Rodriguez-Bano J, Valles J, Palomar M, Tornos P, Bouza E; Sociedad Espanola de Enfermedades Infecciosas y Microbiologia Clinica. [Consensus document for the treatment of bacteremia and endocarditis caused by methicillin-resistent Staphylococcus aureus. Sociedad Espanola de Enfermedades Infecciosas y Microbiologia Clinica]. Enferm Infecc Microbiol Clin. 2009 Feb;27(2):105-15. doi: 10.1016/j.eimc.2008.09.003. Epub 2009 Feb 11. Spanish. PMID 19254641
- [Background] Popovic M, Steinort D, Pillai S, Joukhadar C. Fosfomycin: an old, new friend? Eur J Clin Microbiol Infect Dis. 2010 Feb;29(2):127-42. doi: 10.1007/s10096-009-0833-2. Epub 2009 Nov 14. PMID 19915879
- [Background] Kastoris AC, Rafailidis PI, Vouloumanou EK, Gkegkes ID, Falagas ME. Synergy of fosfomycin with other antibiotics for Gram-positive and Gram-negative bacteria. Eur J Clin Pharmacol. 2010 Apr;66(4):359-68. doi: 10.1007/s00228-010-0794-5. Epub 2010 Feb 26. PMID 20186407
- [Background] Liu C, Bayer A, Cosgrove SE, Daum RS, Fridkin SK, Gorwitz RJ, Kaplan SL, Karchmer AW, Levine DP, Murray BE, J Rybak M, Talan DA, Chambers HF. Clinical practice guidelines by the infectious diseases society of america for the treatment of methicillin-resistant Staphylococcus aureus infections in adults and children: executive summary. Clin Infect Dis. 2011 Feb 1;52(3):285-92. doi: 10.1093/cid/cir034. PMID 21217178
- [Background] Wu G, Abraham T, Rapp J, Vastey F, Saad N, Balmir E. Daptomycin: evaluation of a high-dose treatment strategy. Int J Antimicrob Agents. 2011 Sep;38(3):192-6. doi: 10.1016/j.ijantimicag.2011.03.006. Epub 2011 May 6. PMID 21549573
- [Background] Chen LY, Huang CH, Kuo SC, Hsiao CY, Lin ML, Wang FD, Fung CP. High-dose daptomycin and fosfomycin treatment of a patient with endocarditis caused by daptomycin-nonsusceptible Staphylococcus aureus: case report. BMC Infect Dis. 2011 May 26;11:152. doi: 10.1186/1471-2334-11-152. PMID 21612672
- [Background] Miro JM, Entenza JM, Del Rio A, Velasco M, Castaneda X, Garcia de la Maria C, Giddey M, Armero Y, Pericas JM, Cervera C, Mestres CA, Almela M, Falces C, Marco F, Moreillon P, Moreno A; Hospital Clinic Experimental Endocarditis Study Group. High-dose daptomycin plus fosfomycin is safe and effective in treating methicillin-susceptible and methicillin-resistant Staphylococcus aureus endocarditis. Antimicrob Agents Chemother. 2012 Aug;56(8):4511-5. doi: 10.1128/AAC.06449-11. Epub 2012 May 29. PMID 22644033
- [Background] Kullar R, Davis SL, Levine DP, Zhao JJ, Crank CW, Segreti J, Sakoulas G, Cosgrove SE, Rybak MJ. High-dose daptomycin for treatment of complicated gram-positive infections: a large, multicenter, retrospective study. Pharmacotherapy. 2011 Jun;31(6):527-36. doi: 10.1592/phco.31.6.527. PMID 21923436
- [Background] Gasch O, Ayats J, Angeles Dominguez M, Tubau F, Linares J, Pena C, Grau I, Pallares R, Gudiol F, Ariza J, Pujol M. Epidemiology of methicillin-resistant Staphylococcus aureus (MRSA) bloodstream infection: secular trends over 19 years at a university hospital. Medicine (Baltimore). 2011 Sep;90(5):319-327. doi: 10.1097/MD.0b013e31822f0b54. PMID 21862935
- [Background] Gasch O, Camoez M, Dominguez MA, Padilla B, Pintado V, Almirante B, Molina J, Lopez-Medrano F, Ruiz E, Martinez JA, Bereciartua E, Rodriguez-Lopez F, Fernandez-Mazarrasa C, Goenaga MA, Benito N, Rodriguez-Bano J, Espejo E, Pujol M; REIPI/GEIH Study Groups. Predictive factors for mortality in patients with methicillin-resistant Staphylococcus aureus bloodstream infection: impact on outcome of host, microorganism and therapy. Clin Microbiol Infect. 2013 Nov;19(11):1049-57. doi: 10.1111/1469-0691.12108. Epub 2013 Jan 17. PMID 23331461
- [Background] Garrigos C, Murillo O, Lora-Tamayo J, Verdaguer R, Tubau F, Cabellos C, Cabo J, Ariza J. Fosfomycin-daptomycin and other fosfomycin combinations as alternative therapies in experimental foreign-body infection by methicillin-resistant Staphylococcus aureus. Antimicrob Agents Chemother. 2013 Jan;57(1):606-10. doi: 10.1128/AAC.01570-12. Epub 2012 Oct 22. PMID 23089756
- [Background] Lai CC, Sheng WH, Wang JT, Cheng A, Chuang YC, Chen YC, Chang SC. Safety and efficacy of high-dose daptomycin as salvage therapy for severe gram-positive bacterial sepsis in hospitalized adult patients. BMC Infect Dis. 2013 Feb 4;13:66. doi: 10.1186/1471-2334-13-66. PMID 23379510
- [Derived] Pujol M, Miro JM, Shaw E, Aguado JM, San-Juan R, Puig-Asensio M, Pigrau C, Calbo E, Montejo M, Rodriguez-Alvarez R, Garcia-Pais MJ, Pintado V, Escudero-Sanchez R, Lopez-Contreras J, Morata L, Montero M, Andres M, Pasquau J, Arenas MD, Padilla B, Murillas J, Jover-Saenz A, Lopez-Cortes LE, Garcia-Pardo G, Gasch O, Videla S, Hereu P, Tebe C, Pallares N, Sanllorente M, Dominguez MA, Camara J, Ferrer A, Padulles A, Cuervo G, Carratala J; MRSA Bacteremia (BACSARM) Trial Investigators. Daptomycin Plus Fosfomycin Versus Daptomycin Alone for Methicillin-resistant Staphylococcus aureus Bacteremia and Endocarditis: A Randomized Clinical Trial. Clin Infect Dis. 2021 May 4;72(9):1517-1525. doi: 10.1093/cid/ciaa1081. PMID 32725216
- [Derived] Shaw E, Miro JM, Puig-Asensio M, Pigrau C, Barcenilla F, Murillas J, Garcia-Pardo G, Espejo E, Padilla B, Garcia-Reyne A, Pasquau J, Rodriguez-Bano J, Lopez-Contreras J, Montero M, de la Calle C, Pintado V, Calbo E, Gasch O, Montejo M, Salavert M, Garcia-Pais MJ, Carratala J, Pujol M; Spanish Network for Research in Infectious Diseases (REIPI RD12/0015); Instituto de Salud Carlos III, Madrid, Spain; GEIH (Hospital Infection Study Group). Daptomycin plus fosfomycin versus daptomycin monotherapy in treating MRSA: protocol of a multicentre, randomised, phase III trial. BMJ Open. 2015 Mar 11;5(3):e006723. doi: 10.1136/bmjopen-2014-006723. PMID 25762232